CLINICAL TRIAL: NCT07318675
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HW211026 Ointment After Single or Multiple Doses in Subjects With Actinic Keratosis
Brief Title: A Phase Ib Study of HW211026 Ointment in Patients With Actinic Keratosis.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hubei Bio-Pharmaceutical Industrial Technological Institute Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HW211026-102
Record Dates: First submitted 2025-12-16; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Actinic Keratosis (AK)
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HW211026 (Experimental): Single or multiple topical doses of HW211026
  Interventions: Drug: HW211026
- Placebo (Placebo Comparator): Single or multiple topical doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HW211026 — Dose 1 and Dose 2
  Arms: HW211026
Drug: Placebo — Dose 1 and Dose 2
  Arms: Placebo

SUMMARY:
This is a phase Ib study to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) characteristics of HW211026 ointment after single or multiple topical administrations in patients with actinic keratosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed as actinic keratosis by histopathology, with Olsen grade 1 or 2.
* A 100 cm² treatment field can be demarcated on the face, which covers clinically typical actinic keratosis lesions (excluding lesions on the lips, perioral region, eyelids, periorbital area, inside and around the nostrils, and the inner ear canal).
* Willing to avoid direct exposure of the treatment field to sunlight or ultraviolet (UV) radiation during the study.

Key Exclusion Criteria:

* Subjects with any of the following conditions within the treatment field：

  * Presence of clinically atypical and/or rapidly changing actinic keratosis lesions, such as hypertrophic lesions, hyperkeratotic lesions, and/or cutaneous horns;
  * Maximum diameter of a single lesion > 2 cm；
  * History of invasive squamous cell carcinoma, Bowen's disease, basal cell carcinoma, or other malignant tumors；
  * Presence of other skin diseases or conditions that may cause difficulties in examination or evaluation.
* treatment field falls within any of the following locations:

  * Presence of incompletely healed wounds within a 5 cm radius of the treatment field;
  * Presence of suspected squamous cell carcinoma, basal cell carcinoma, or other tumors within a 5 cm radius of the treatment field.
* Subjects with other skin diseases (e.g., atopic dermatitis, psoriasis, eczema, etc.) or other skin conditions (e.g., tattoos, birthmarks, ulcerations, scars, open wounds, etc.) that the investigator deems may interfere with the assessment of safety or efficacy.
* Subjects with severe cardiovascular and cerebrovascular diseases.
* Receipt of any systemic drug therapy for actinic keratosis within 6 months prior to screening.
* Receipt of any topical intervention for actinic keratosis on the administration area within 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | up to 28 days
  To assess the safety and tolerability of single or multiple topical doses of HW211026 in adults with actinic keratosis

SECONDARY OUTCOMES:
The maximum serum concentration(Cmax) | up to 10 days
  PK Parameter
The Area Under the Curve from dosing to the time of the last measured concentration | up to 10 days
  PK Parameter
The time to reach Cmax(Tmax) | up to 10 days
  PK Parameter
The Half life(t1/2) | up to 10 days
  PK Parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No